CLINICAL TRIAL: NCT04448327
Title: Sex-Dependent Impact of Transcutaneous Vagal Nerve Stimulation on the Stress Response Circuitry and Autonomic Dysregulation in Major Depression
Brief Title: Impact of Transcutaneous Vagal Nerve Stimulation on Stress Response in Major Depression
Acronym: tVNS_MDD_Sex
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ronald Garcia, Instructor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020P001212; 1U54MH118919-01A1 (NIH)
Record Dates: First submitted 2020-06-17; First posted 2020-06-25 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Major Depressive Disorder
Keywords: Autonomic Nervous System; Transcutaneous Vagus Nerve Stimulation; Stress Response Circuitry; Functional Magnetic Resonance Imaging; Sex Differences
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Active tVNS (Experimental): Expiratory-gated transcutaneous vagus nerve stimulation on the left auricle
  Interventions: Device: active tVNS
- Sham tVNS (Sham Comparator): Sham transcutaneous vagus nerve stimulation on the left auricle
  Interventions: Device: Sham tVNS

INTERVENTIONS:
Device: active tVNS — non-painful electrical stimulation of the auricle for 30 minutes during a functional magnetic resonance imaging session
  Other Names: transcutaneous vagus nerve stimulation
  Arms: Active tVNS
Device: Sham tVNS — Sham stimulation of the auricle for 30 minutes during a functional magnetic resonance imaging session
  Other Names: transcutaneous vagus nerve stimulation
  Arms: Sham tVNS

SUMMARY:
This study will identify the sex-dependent impact of expiratory-gated transcutaneous vagus nerve stimulation (tVNS) on the modulation of the stress response circuitry and associated physiology in major depressive disorder (MDD). We will evaluate a sample of 80 adults with recurrent MDD randomized to receive active or sham expiratory-gated tVNS during a functional magnetic resonance imaging (fMRI) session, with simultaneous mood and physiological assessments. We hypothesize that expiratory-gated tVNS will effectively modulate, in a sex-dependent manner, specific brainstem-cortical pathways of the stress circuitry and attenuate physiological deficits in MDD.

DETAILED DESCRIPTION:
Major depressive disorder (MDD) is a leading cause of morbidity and disability worldwide with abnormalities in the stress response circuitry and central autonomic network. Many of these regions are sexually dimorphic and related with sex differences in mood and hypothalamic-pituitary-adrenal (HPA) axis modulation, the dysregulation of which is associated with alterations of hormone and immune responses to stress, autonomic dysfunction and increased cardiovascular risk. The primary goal of this study is to use non-invasive neuromodulatory stimulation of the vagus to target the circuitry associated with stress-immune function and map its neuroanatomic and physiological effects in MDD by sex. Vagal nerve stimulation (VNS), FDA-approved for MDD, modulates brain circuitry implicated in mood/anxiety and autonomic regulation, however, it is implanted and thus invasive. We propose the use of a physiologically-enhanced transcutaneous VNS (tVNS) as a low risk, non-invasive, and inexpensive alternative. While tVNS has had beneficial effects on depressive symptomatology and autonomic regulation, current stimulation parameters are based on historical iVNS data that included mostly male populations. We propose that tVNS effects on the regulation of specific brainstem-cortical pathways is modulated by sex. Moreover, as the dorsal medullary vagal system operates in tune with respiration, we recently demonstrated that tVNS can be optimized by gating stimulation to respiration. Thus, this study proposes to identify the sex-dependent impact of expiratory-gated tVNS on the modulation of stress response circuitry alterations and physiological dysregulation of recurrent MDD. We will evaluate a sample of 80 adults with recurrent MDD randomized to receive active tVNS or sham stimulation during a functional magnetic resonance imaging (fMRI) session. The fMRI session will include a stress challenge designed to elicit a sympatho-excitatory state, with simultaneous mood and physiological assessments, including hormonal and dynamic cardiovagal heart rate variability (HRV) evaluations. We hypothesize that expiratory-gated tVNS will effectively modulate specific brainstem-cortical pathways of the stress response circuitry and will attenuate physiological deficits of recurrent MDD patients. We further hypothesize that tVNS will impact brain activity and physiology in sex-dependent ways.

ELIGIBILITY:
Inclusion Criteria:

* Current or past diagnosis of recurrent Major Depressive Disorder

Exclusion Criteria:

* History of neuroleptic use
* Any psychiatric disorder involving a history of psychosis (e.g. schizophrenia, bipolar I disorder)
* Active suicidal ideation with intent and/or plan or history of a suicide attempt within the last year
* Moderate or severe substance use disorder within the past 12 months
* Diagnosis of significant cardiovascular or cerebrovascular disease (e.g. congestive heart failure, stroke, cardiac conduction disorders, history of asystole or non-sustained ventricular tachycardia)
* Diseases affecting the CNS (e.g. MS, epilepsy, neurodegenerative diseases, etc.)
* Traumatic brain injury with cognitive sequelae
* MRI or tVNS contraindications (e.g. claustrophobia, metallic implants or devices)
* Pregnancy (uncommon, given the age of this cohort is 50+ years) due to unknown health risks for the fetus

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-01-29 (Actual); Primary Completion 2025-06-13 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Brain activity during functional magnetic resonance imaging (fMRI) | 1 hour
  Changes in fMRI BOLD signal (percent BOLD signal change) of the stress response circuitry between active and sham tVNS.
Cardiac autonomic function during functional magnetic resonance imaging (fMRI) | 1 hour
  Changes in cardiac autonomic function (High Frequency power-Heart Rate Variability) between active and sham tVNS.

SECONDARY OUTCOMES:
Change in serum cortisol levels | 2 hours
  Changes in serum cortisol levels from baseline to post-stimulation will be assessed and compared between active and sham tVNS
Change in serum levels of pro-inflammatory cytokines | 2 hours
  Changes in serum levels of proinflammatory cytokines (IL1B, IL6, TNF alfa) from baseline to post-stimulation will be assessed and compared between active and sham tVNS
Change in depressive symptoms assessed by the Beck Depression Inventory | 2 hours
  Changes from baseline to post-stimulation in the score of the Beck Depression Inventory will be compared between active and sham tVNS. (Beck depression inventory minimum score= 0, maximum score= 63; higher total scores indicate more severe depressive symptoms)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Garcia, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No